CLINICAL TRIAL: NCT03853044
Title: A Phase 2, Open-Label Study to Evaluate the Safety and Efficacy of Chidamide Combined With CHOP(Cyclophosphamide, Doxorubicin, Vincristine, Prednisone ) in Untreated Subjects With Angioimmunoblastic T Cell Lymphoma
Brief Title: Study Evaluating the Safety and Efficacy of C-CHOP in Untreated Subjects With Angioimmunoblastic T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-CHOP
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Angioimmunoblastic T-cell Lymphoma
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide plus CHOP (Experimental): Participants received six 21-day cycles of chidamide, combined with six cycles of standard cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) chemotherapy (21-day cycles).
  Interventions: Drug: Chidamide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Chidamide — Chidamide 20mg per day administered orally on Day 1, 4, 8, 11 of each 21-day cycle for 6 cycles
Drug: Cyclophosphamide — Cyclophosphamide 750 milligrams per square metre (mg/m^2), administered intravenously (IV) on Day 1 of each 21-day cycle.
Drug: Doxorubicin — Doxorubicin 50 mg/m^2 IV, administered on Day 1 of each 21-day cycle.
Drug: Vincristine — Vincristine 1.4 mg/m^2 (maximum 2 mg) IV, administered on Day 1 of each 21-day cycle.
Drug: Prednisone — Prednisone 60mg/m2 , Maximum 100 mg , (or equivalent prednisolone or methylprednisolone), administered orally on Days 1-5 of each 21-day cycle.

SUMMARY:
This is a single-arm, open-label phase 2study of Chidamide in combination with CHOP in the treatment of subjects with untreated angioimmunoblastic T cell lymphoma.

DETAILED DESCRIPTION:
This open-label, single arm study will evaluate the efficacy and safety of chidamide in combination with cyclophosphamide, doxorubicin, vincristine, and prednisolone or prednisone (CHOP) chemotherapy in previously untreated subjects with angioimmunoblastic T cell lymphoma. Subjects will receive 6 cycles of Chidamide 20mg, day 1,4,8,11, orally (PO) every 21 days, in addition to 6 cycles of CHOP chemotherapy IV every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed angioimmunoblastic T cell lymphoma
2. Treatment naive
3. Age > 18 years
4. Must has measurable lesion in CT or PET-CT prior to treatment
5. ECOG 0,1,2
6. Informed consented

Exclusion Criteria:

1. Has accepted Chemotherapy before
2. Has accepted autologous Stem cell transplantation before
3. History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix 3 years prior to study treatment
4. Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
5. Primary CNS lymphoma
6. LVEF≤50%
7. Lab at enrollment (Unless caused by lymphoma): Neutrophile<1.5*10^9/L ;Platelet<75*10^9/L; ALT or AST >2*ULN; AKP or bilirubin >1.5*ULN ;Creatinine>1.5*ULN
8. Other uncontrollable medical condition that may that may interfere the participation of the study
9. Not able to comply to the protocol for mental or other unknown reasons
10. Pregnant or lactation
11. HIV infection
12. If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA,DNA positive patients cannot be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2018-12-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Overall response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with response(complete response and partial response) was determined on the basis of investigator assessments according to 2014 Lugano criteria
Progression free survival | Baseline up to data cut-off (up to approximately 4 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival in the overall study population was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event.
Duration of response | Baseline up to data cut-off (up to approximately 4 years)
  time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Baseline up to data cut-off (up to approximately 4 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Core 30 (EORTC QLQ-C30) Domain Scores | Baseline (pre-dose [Hour 0] on Cycle1 Day1), Cycle3 Day 1, end of treatment (up to Month 6), every 3 months 1st year, every 6 months 2nd year, and 12 months thereafter up to data cut-off, up to approximately 4 years (cycle length = 21 days) ]
  The EORTC QLQ-C30 is a health-related quality of life questionnaire. A higher score indicates better quality of life, with changes of 5 to 10 points considered to be a minimally important difference to participants.

OTHER OUTCOMES:
Circulating free Deoxyribonucleic Acid (cfDNA) monitoring | Baseline up to data cut-off (up to approximately 4 years)
  cfDNA in peripheral blood assessed by local lab

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD. PhD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No